CLINICAL TRIAL: NCT04280965
Title: Quetiapine Augmentation of Prolonged Exposure (PE) Therapy for the Treatment of Co-occurring PTSD and Mild Traumatic Brain Injury
Brief Title: Quetiapine Augmentation of PE Therapy for the Treatment of Co-occurring PTSD and Mild Traumatic Brain Injury
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Central MIRECC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-200H
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quetiapine (Experimental): Flexible dosing begins at 50 mg, titrating up to 100 mg at the end of week 2 with additional doses up to 400 mg per day if needed
  Interventions: Drug: Quetiapine Fumarate
- Treatment As Usual (TAU) (Active Comparator): Standard of care medications
  Interventions: Other: Standard of care meducations

INTERVENTIONS:
Drug: Quetiapine Fumarate — Atypical antipsychotic
  Other Names: Seroquel
  Arms: Quetiapine
Other: Standard of care meducations — SSRI's/SNRI's/Trazodone/Prazosin/Hydroxyzine
  Arms: Treatment As Usual (TAU)

SUMMARY:
A pilot study to evaluate feasibility for a full-scale merit application. Specifically, for veterans considering prolonged exposure (PE) therapy, following the model established by Foa et al, we need to establish safety, and feasibility of quetiapine compared to treatment as usual (TAU) which employs multiple medications commonly used for PTSD in the VA system.

ELIGIBILITY:
Inclusion Criteria:

1. All treatment seeking adult (≥ 18 years)
2. Veterans with mTBI who meet PTSD diagnosis and have a CAPS-5 score of 25 or greater. Diagnosis will be determined using the provisional PTSD diagnosis convention recommended by the National Center of PTSD which requires at least moderate ratings (2 or more) on at least 1 B item (items #1-5), 1 C item (items #6-7), 2 D items (#8-14), and 2 E items (items #15-20) of the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).

Exclusion Criteria: (1) Pregnant or lactating women and those of child-bearing potential not using a reliable method of contraception; (2) Individuals meeting DSM-5 criteria for schizophrenia, schizoaffective disorder, or neurocognitive disorder; (3) Individuals currently taking any typical or atypical antipsychotic medication or individuals using daily benzodiazepines including nonbenzodiazepine z-drugs for sleep as they have effects similar to benzodiazepines for sleep. (Note: benzodiazepine use is contraindicated as they may impair learning required for progress with PE) (4) Individuals with known intolerance to quetiapine or a history of clinically unstable heart, lung, liver, renal or endocrinological condition, diabetes mellitus, and/or seizure disorder. (5) Individuals with substance use disorder severe enough to require medical detoxification.

(6) Individuals who report suicidal or homicidal ideations in the past month severe enough to warrant inpatient admission.

(7) Individuals with current or known history of cardiac arrhythmia or QTc interval ≥ 450 milliseconds. (Note) Patients requiring other anti-arousal medication for general medical conditions such as antihypertensive medications, beta blockers etc., for hypertension, anti-thyroid medications for hyperthyroidism, and/or anti-epileptic medications, divalproex, levetiracetam, or carbamazepine for seizure disorder may be included if stable for at least 1 month before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Percentage compliance in completing PE sessions | 1.5 yr
  The percentage of participants who complete the 10 sessions of Prolonged Exposure (PE) within 12-14 weeks of beginning treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Baig, MD, Principal Investigator — South Texas Veterans Health Care System
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD that underlie results in publication
Supporting Information: SAP
Time Frame: Anticipated June 2023
Access Criteria: Acceptance for publication by journal

REFERENCES:
- [Derived] Baig MR, Beck RD, Wilson JL, Lemmer JA, Meraj A, Meyer EC, Mintz J, Peterson AL, Roache JD. Quetiapine augmentation of prolonged exposure therapy in veterans with PTSD and a history of mild traumatic brain injury: design and methodology of a pilot study. Mil Med Res. 2020 Oct 8;7(1):46. doi: 10.1186/s40779-020-00278-0. PMID 33032657